CLINICAL TRIAL: NCT02097953
Title: Influence of Rifampin Co-Administration on the Pharmacokinetic Profile of Daptomycin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Principal Investigator, Russell Benefield, Pharmacist, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00069136
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Drug Interactions; Pharmacokinetics
Keywords: Daptomycin; Rifampin; P-glycoprotein; Pharmacokinetic
MeSH Terms: interventions — Daptomycin; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daptomycin and Rifampin (Experimental): Drug: Daptomycin Daptomycin 6 mg/kg will be given by IV infusion on the first study day Drug: Rifampin Rifampin 600 mg capsules will be given orally once daily for 14 days starting on study day 2 Drug: Daptomycin Daptomycin 6 mg/kg will be given by IV infusion on study day 15
  Interventions: Drug: Daptomycin; Drug: Rifampin

INTERVENTIONS:
Drug: Daptomycin
  Other Names: Cubicin
Drug: Rifampin
  Other Names: Rifadin

SUMMARY:
The purpose of this study is to understand how an antibiotic, rifampin, may change the blood levels of another antibiotic, daptomycin, in the body. In addition, the effect of polymorphisms in P-glycoprotein (a protein involved in the removal of daptomycin from the body) on the blood levels of daptomycin will be evaluated. The hypotheses are that rifampin will decrease the blood levels of daptomycin and that the effect will be greater for certain P-glycoprotein polymorphisms.

DETAILED DESCRIPTION:
This will be an open-label, sequential pharmacokinetic study in 12 healthy volunteers. After providing informed consent, participants meeting inclusion criteria will be administered daptomycin 6 mg/kg over 2 minutes and blood and urine samples will be collected over a 24 hour period after infusion. Following this, participants will be given a 13 day supply of rifampin 600 mg/day to be taken at home. After completion of the rifampin course, a second pharmacokinetic sampling will be performed (day 15 overall). Participants will be administered a dose of rifampin 600 mg then once again be administered daptomycin 6 mg/kg over 2 minutes and blood and urine samples will be collected over a second 24 hour period. A blood sample will be obtained at the first study visit for determination of each participant's P-glycoprotein genotype.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* If female of child bearing potential, on reliable method of contraception and negative pregnancy test at enrollment

Exclusion Criteria:

* Obesity (body mass index > 30)
* Creatinine clearance < 80 ml/min
* Creatine phosphokinase > 2 times upper limit of normal at enrollment
* Aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase > 3 times upper limit of normal at enrollment
* History of liver disease or cirrhosis
* History of congestive heart failure
* Allergy or intolerance to rifampin or daptomycin
* Need for concomitant non-study medications during the study period
* Inability to abstain from grapefruit juice or herbal supplements (such as St. John's wort) during the study period
* Receipt of study drugs within 30 days prior to enrollment
* Pregnancy or lactation
* Inability to adhere to study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Daptomycin total, renal, and non-renal clearance | 14 days
  Total, renal, and non-renal clearance of daptomycin before and after administration of rifampin
Daptomycin Volume of Distribution | 14 days
  The volume of distribution of daptomycin before and after administration of rifampin
Daptomycin Elimination Rate Constant | 14 days
  The elimination rate constant of daptomycin before and after administration of rifampin
Daptomycin Free and Total Peak Concentrations | 14 days
  The free and total peak concentrations of daptomycin before and after administration of rifampin
Daptomycin Free and Total 24 hour Concentrations | 14 days
  The free and total 24 hour concentrations of daptomycin before and after administration of rifampin
Daptomycin Free and Total Area Under the Concentration-Time Curve (AUC) from 0 to 24 hours | 14 days
  The free and total AUC from 0 to 24 hours of daptomycin before and after administration of rifampin
Daptomycin Free and Total AUC from 0 to Infinity | 14 days
  The free and total AUC from 0 to infinity of daptomycin before and after administration of rifampin
Percent Protein Binding of Daptomycin | 14 days
  The percent protein binding of daptomycin before and after administration of rifampin

SECONDARY OUTCOMES:
P-glycoprotein Polymorphism | 14 days
  The effect of different P-glycoprotein polymorphisms on the pharmacokinetic profile of daptomycin before and after administration of rifampin will be assessed
Number of Participants with Adverse Events | 45 days
  Safety monitoring will be done by regular adverse event assessment, laboratory and vital sign monitoring, and physical exam.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Benefield, Pharm.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States